CLINICAL TRIAL: NCT01501214
Title: A Randomized Double Blind Comparison of Atosiban in Patients Undergoing in Vitro Fertilization Treatment
Brief Title: Use of Atosiban in in Vitro Fertilization (IVF) Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Vietnam National University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKUQMHCARE001
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Subfertility
Keywords: atosiban; in vitro fertilization; subfertility
MeSH Terms: conditions — Infertility | interventions — atosiban; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atosiban (Active Comparator)
  Interventions: Drug: Atosiban
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Atosiban — Patients in the atosiban group will receive intravenous atosiban 30 min before the transfer with a bolus dose of 6.75 mg, and the infusion will be continued with an infusion rate of 18 mg/h. After performing ET, the dose of atosiban will be reduced to 6 mg/h and the infusion will be continued for 2 hours (total administered dose: 37.5 mg). Those in the placebo group will receive normal saline only.
  Other Names: Tractocile
  Arms: Atosiban
Drug: Normal saline — Normal saline given
  Arms: Placebo

SUMMARY:
The hypothesis of this randomized double blind study is that the live birth rates are significantly higher after the use of atosiban prior to the embryo transfer in patients undergoing in vitro fertilization (IVF) treatment. This study aims to compare the live birth rates of IVF treatment between patients receiving atosiban and placebo prior to the transfer.

DETAILED DESCRIPTION:
In-vitro fertilization-embryo transfer (IVF-ET) treatment involves multiple follicular development following ovarian stimulation, oocyte retrieval and ET after fertilization. Despite recent advances in ovarian stimulation, the method of assisted fertilization and improved culture conditions, the implantation potential of embryos remains around 20-25% for a long time.

ET is the final step of an IVF cycle and its success depends on the embryo quality, the endometrial receptivity and uterine contractions. Uterine contractions play an important role in embryo implantation (Fanchin, 2009) as excessive uterine contractions may expel embryos from the uterus and decrease the implantation potential of embryos (Fanchin et al., 1998).

Ovarian stimulation is used in the great majority of IVF programs so that multiple embryos are available for selection and transfer. However, supraphysiological concentrations of oestradiol following ovarian stimulation may induce endometrial production of oxytocin, formation of oxytocin receptors, and indirectly formation/release of PGF2a (Richter et al., 2004; Liedman et al., 2008). It has been shown that uterine contractile activity in IVF cycles is increased by approximately 6-fold when measured before ET as compared with the situation before ovulation in the natural cycle (Ayoubi et al., 2003). Fanchin et al. (1998) have estimated that about 30% of patients undergoing ET have pronounced uterine contractions. Uterine contractions can also be triggered after excessive cervical manipulation in difficult transfer procedure (Fanchin et al., 1998).

Drugs to inhibit increased uterine contractions at the time of ET are an attractive approach to improve the IVF success. However, the use of beta agonists or non-steroid anti-inflammatory drugs has not been shown to provide sufficient benefit (Bernabeu et al., 2006; Moon et al., 2004; Tsirigotis et al., 2000). Uterine contractions involve oxytocin and therefore inhibition of oxytocin receptors may improve the IVF success by decreasing uterine contractions, interfering with PGF2a/oxytocin systems and possibly improving endometrial perfusion (Vedernikov et al., 2006).

Atosiban, a combined oxytocin/vasopressin V1A antagonist, is currently registered for clinical use in women suffering from preterm labour. In a multicentre, randomized, placebo-controlled trial, it has been shown to reduce the frequency and amplitude of uterine contractions in egg donors when compared with placebo (Blockeel et al., 2009; Pierson et al., 2009; Visnova et al., 2009). There was a lack of an embryotoxic effect of atosiban in concentrations up to 50-fold therapeutic blood concentrations (Pierzynski et al., 2007). Atosiban did not affect the survival of 1-cell rabbit embryos, nor decrease the percentage of hatched rabbit blastocysts. The human sperm motility bioassay also showed no adverse influence.

ELIGIBILITY:
Inclusion Criteria:

* Age < 43 years
* Normal uterine cavity shown on ultrasound scanning

Exclusion Criteria:

* Age >=43
* Three previous IVF cycles
* Use of donor oocytes
* Natural IVF or IVM cycles
* Abnormal uterine cavity on ultrasound scanning
* ET canceled because of absent fertilization or risk of ovarian hyperstimulation syndrome
* Blastocyst transfer
* Undergoing preimplantation genetic diagnosis
* Recruited in the same study before

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
live birth rate | 9 months

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — The University of Hong Kong
Locations (2):
- Reproductive Medical Center of Nanfang Hospital, Guangzhou, Guangdong, China
- CGRH, School of Medicine, Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Ayoubi JM, Epiney M, Brioschi PA, Fanchin R, Chardonnens D, de Ziegler D. Comparison of changes in uterine contraction frequency after ovulation in the menstrual cycle and in in vitro fertilization cycles. Fertil Steril. 2003 May;79(5):1101-5. doi: 10.1016/s0015-0282(03)00179-1. PMID 12738502
- [Background] Bernabeu R, Roca M, Torres A, Ten J. Indomethacin effect on implantation rates in oocyte recipients. Hum Reprod. 2006 Feb;21(2):364-9. doi: 10.1093/humrep/dei343. Epub 2005 Nov 10. PMID 16284067
- [Background] Blockeel C, Pierson R, Popovic-Todorovic B, Visnova HA, Garcı´a-Velasco HA, Mra´zek M, Barri PN, Pierzynski P, Kuczynski W, Devroey P, Breinholt V, Erichsen L, Klein BM, Arce JC. Effects of barusiban and atosiban on frequency of uterine contractions in the luteal phase after stimulation: a randomized placebo controlled trial. Hum. Reprod. 24 (Suppl. 1), i26, 2009.
- [Background] Fanchin R, Ayoubi JM. Uterine dynamics: impact on the human reproduction process. Reprod Biomed Online. 2009;18 Suppl 2:57-62. doi: 10.1016/s1472-6483(10)60450-6. PMID 19406033
- [Background] Fanchin R, Righini C, Olivennes F, Taylor S, de Ziegler D, Frydman R. Uterine contractions at the time of embryo transfer alter pregnancy rates after in-vitro fertilization. Hum Reprod. 1998 Jul;13(7):1968-74. doi: 10.1093/humrep/13.7.1968. PMID 9740459
- [Background] Liedman R, Hansson SR, Howe D, Igidbashian S, McLeod A, Russell RJ, Akerlund M. Reproductive hormones in plasma over the menstrual cycle in primary dysmenorrhea compared with healthy subjects. Gynecol Endocrinol. 2008 Sep;24(9):508-13. doi: 10.1080/09513590802306218. PMID 18958771
- [Background] Moon HS, Park SH, Lee JO, Kim KS, Joo BS. Treatment with piroxicam before embryo transfer increases the pregnancy rate after in vitro fertilization and embryo transfer. Fertil Steril. 2004 Oct;82(4):816-20. doi: 10.1016/j.fertnstert.2004.02.140. PMID 15482753
- [Background] Pierson R, Deptuch JJ, Invik J, Klein BM, Breinholt V, Arce JC. Reproducibility of uterine contractility assessments based on transvaginal ultrasound cine-loop recordings. Hum. Reprod. 24 (Suppl. 1), i103, 2009.
- [Background] Pierzynski P, Gajda B, Smorag Z, Rasmussen AD, Kuczynski W. Effect of atosiban on rabbit embryo development and human sperm motility. Fertil Steril. 2007 May;87(5):1147-52. doi: 10.1016/j.fertnstert.2006.08.089. Epub 2007 Jan 16. PMID 17224148
- [Background] Richter ON, Kubler K, Schmolling J, Kupka M, Reinsberg J, Ulrich U, van der Ven H, Wardelmann E, van der Ven K. Oxytocin receptor gene expression of estrogen-stimulated human myometrium in extracorporeally perfused non-pregnant uteri. Mol Hum Reprod. 2004 May;10(5):339-46. doi: 10.1093/molehr/gah039. Epub 2004 Mar 25. PMID 15044599
- [Background] Tsirigotis M, Pelekanos M, Gilhespie S, Gregorakis S, Pistofidis G. Ritodrine use during the peri-implantation period reduces uterine contractility and improves implantation and pregnancy rates post-ivf. Hum. Reprod. 15, (Abs. Bk 1), O-024, 10, 2000.
- [Background] Vedernikov Y, Betancourt A, Shi S, Shi L, Reinheimer T, Garfield R. (2006) Oxytocin antagonistic effect of barusiban and atosiban in isolated uterine artery from late pregnant rats. In: Annual scientific meeting of the Society for Gynecologic Investigation. Toronto, Canada.
- [Background] Visnova H, Coroleu B, Piro M, Blockeel C, Mrazek M, Arce JC. Barusiban and atosiban for reduction of uterine contractions on day of embryo transfer do not alter the endocrine profile at time of implantation. Hum. Reprod. 24 (Suppl. 1), i178, 2009.
- [Derived] Ng EH, Li RH, Chen L, Lan VT, Tuong HM, Quan S. A randomized double blind comparison of atosiban in patients undergoing IVF treatment. Hum Reprod. 2014 Dec;29(12):2687-94. doi: 10.1093/humrep/deu263. Epub 2014 Oct 21. PMID 25336707